CLINICAL TRIAL: NCT05628207
Title: Evaluation of the SCALED (SCaling AcceptabLE cDs) Approach for the Implementation of Interoperable CDS for Venous Thromboembolism Prevention - CDS Data
Brief Title: Evaluation of the SCALED (SCaling AcceptabLE cDs)
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: HRP-595
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury; Venous Thromboembolism
MeSH Terms: conditions — Brain Injuries, Traumatic; Venous Thromboembolism | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 4 hospitals using CDS TBI: healthcare system leveraging the rigorous approach, SCALED (SCaling AcceptabLE cDs), to guide CDS scaling across the system in VTE prevention.
  Interventions: Other: Observational
- 3 hospitals not using CDS TBI (control): healthcare system not leveraging the rigorous approach, SCALED (SCaling AcceptabLE cDs), to guide CDS scaling across the system in VTE prevention.
  Interventions: Other: Observational-control

INTERVENTIONS:
Other: Observational — There is no intervention, the hospitals will adopt a CDS system which prompts users to follow best practice guidelines.
  Groups: 4 hospitals using CDS TBI
Other: Observational-control — There is no intervention, the hospitals will not use the CDS system.
  Groups: 3 hospitals not using CDS TBI (control)

SUMMARY:
This project will adapt a currently deployed Clinical Decision Support (CDS) system to deliver a VTE prevention guideline for adult patients with traumatic brain injury (TBI). We believe this is an ideal PCOR use case given PCORI's continued effort to combat VTE in trauma and our experience previously implementing this guideline. The Our overall goal is to successfully scale, evaluate, and maintain an interoperable TBI CDS across 7 total institutions.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and older
* admitted with a TBI

Exclusion Criteria:

* Patients who die within 24 hours of hospital admission and patients documented as "comfort cares" during the first 72 hours of hospitalization or with mild TBI will be excluded from final analysis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients age 18 and older admitted with a TBI will be eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
primary effectiveness outcome | 2 years and a half
  VTE event rate
Evaluate implementation strategy guided by the EPIS Implementation | 2 years and a half
  the number of patients that received treatment according to the best practice guideline and the % adherence to the guideline per site

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Tignanelli CJ, Shah S, Vock D, Siegel L, Serrano C, Haut E, Switzer S, Martin CL, Rizvi R, Peta V, Jenkins PC, Lemke N, Thyvalikakath T, Osheroff JA, Torres D, Vawdrey D, Callcut RA, Butler M, Melton GB. A pragmatic, stepped-wedge, hybrid type II trial of interoperable clinical decision support to improve venous thromboembolism prophylaxis for patients with traumatic brain injury. Implement Sci. 2024 Aug 5;19(1):57. doi: 10.1186/s13012-024-01386-4. PMID 39103955